CLINICAL TRIAL: NCT04546659
Title: Effects of Retro-walking on Pain, Functional Disability and Performance in Knee Osteoarthritis
Brief Title: Retro-walking in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/1055 Saira Shabbir
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; knee joint; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Osteoarthritic patient receiving Conventional therapy and Retrowalking
  Interventions: Other: Retrowalking; Other: Conventional Therapy
- Group B (Active Comparator): Osteoarthritic patient receiving Conventional therapy
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Retrowalking — Treatment of retro-walking including supervised 10 min retro-walking training with 5 min of warm-up and cool down on a flat surface at their comfortable speed
  Arms: Group A
Other: Conventional Therapy — Treatment of conventional therapy involve Isometric Quadriceps exercise, SLR, Isometric hip adduction exercises, Terminal knee extension exercise 1 set of 10 Reps twice a day.

SUMMARY:
In osteoarthritis the most affected joint is knee due to degenerative changes. Degenerative changes cause age-related wear-and-tear and may be accelerated by injury, health and lifestyle factors, and possibly by genetic predisposition to joint pain or musculoskeletal disorders. Knee osteoarthritis causes pain, swelling & stiffness in joint. Patients unable to perform ADL's and IADL's due to pain.

Various treatment methods are used for management of knee osteoarthritis. But physiotherapy approach is best option for making patients independent after medical management. This study will be a randomized control trial, used to compare the effectiveness of retro-walking and conventional therapy to improve pain, functional disability and performance in knee osteoarthritic patient. Subjects with knee osteoarthritis meeting the predetermined inclusion & exclusion criteria will divide into two groups using lottery method. Time up & Go (TUG), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) & Numeric Pain Rating Scale (NPRS) tools for screening will be used for data collection. Subjects in one group will be treated with retro-walking & conventional therapy and other will be treated with conventional therapy. Each subject will receive a total 6 weeks treatment session, with 3 treatment sessions per week. Recorded values will be analyzed for any change using SPSS 21 version.

DETAILED DESCRIPTION:
Knee osteoarthritis causes chronic disability in the older population worldwide. Its prevalence increases dramatically with age. Prevalence of radiographic osteoarthritis is estimated at 80 % of all adults at or over the age of 65 years. The common impairments such as knee pain, decreased functional mobility, quadriceps strength, and stiffness leading to physical disability have been associated with knee osteoarthritis .

The prevalence of osteoarthritis is gradually in- creasing in both low- and high-income countries.The Global Burden of Disease studies recently indicated that knee osteoarthritis is the fastest increasing major health dis- order and the second global cause of disability. In the lower extremity, the knee is often affected, and knee osteoarthritis results in significant mobility restrictions and a substantial financial burden. The risk of osteoarthritis associated disability is equal to that of cardiac disorders and more common than any other medical problem in older populations. The common clinical manifestations of knee osteoarthritis include pain, stiffness, joint enlargement, crepitus, muscle weakness, deformity, impaired proprioception, reduced joint motion, and disability. Therapeutic exercises are often used to improve physiological impairments such as reduced joint motion, muscle weakness, impaired balance, disability, and proprioception.

Forward walking provides an increased opportunity to train the entire gait cycle, facilitating an enhanced gait pattern in children with cerebral palsy. Backward walking is recommended to improve the components of forward walking in those children. Hoog kamer et al. reported that backward walking uses the same rhythm circuitry of forward walking, but additionally requires specialized control circuits. Gait rehabilitation with backward walking puts emphasis on positioning the foot behind the body and, thus, facilitates hip extension while performing a knee flexion that can be useful for patients who have synergistic influences in the lower extremity. A longer period of muscles activity of the legs during backward walking training can result in greater muscle strength gain as compared with for- ward walking training. Furthermore, training in backward walking could require higher physiological and perceptual responses than forward walking at matched speed, as backward walking is the performance of a novel task for most children with cerebral palsy.

Among the current possible gait training methods, backward walking has emerged as an important therapy. Backward walking is regulated by the same central pattern generator as forward walking. Unlike forward walking, backward walking has no heel contact in the early stance phase and thus leads to lower compression force at the patella femoral joint and decreased force absorption at the knee joint. In addition, lower limb muscle activity during backward walking is intensified on account of the higher recruitment of motor units. During the loading response phase of backward walking, the ground reaction force rapidly increases to support the weight of the entire body. The absence of visual cues during backward walking results in increased spatial and smaller temporal gait parameters. Therefore, backward walking can be considered as a treatment strategy to improve gait.

Many pharmacological treatment strategies may improve disease-related impairments; however, have limited impact on gait. In recent years, backward walking has become an attractive alternative for training and rehabilitation purposes to improve mobility. For individuals with stroke, both over ground and treadmill backward walking training has been affective to improve walking speed, stride length , gait asymmetry, gait cycle phases, functional capacity and balance. Similarly, in children with cerebral palsy, Backward Walking treadmill training improved gait speed, step length, Stride Length and functional capacity and the addition of over ground Backward Walking to a traditional physical therapy program improved overall postural instability.

To our knowledge, there is a lack of studies has evaluated the Effects of Retro-walking on pain, functional disability and performance in knee osteoarthritis. Investigator developed a program to apply retro-walking to Osteoarthritic patients. Repetition of movements will be added to program. This program is design to improve knee performance, functional ability & reduce pain. The purpose of the present study is to examine the efficiency of retro-walking to improve functional disability and performance and reduce pain in patients with osteoarthritis.

Investigator predict that retro-walking will improve performance, functional disability & pain in patients with knee osteoarthritis; they will enhance their performance, movement as well as functional abilities. Also so there is awareness in community for the efficacy of neurodevelopmental therapy for the management in Down syndrome infants.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering with Osteoarthritis knee for three months at least
* Age ranges from 40-70
* knee OA as per the American College of Rheumatology clinical and radiographic diagnostic criteria will participate
* 1-3 radiographic grades on the Kellgren-Lawrence scale
* Both genders will be included
* being able to cooperate
* Bilateral knee osteoarthritis

Exclusion Criteria:

* Traumatic knee pain, fractures or ruptured ligaments, meniscopathy of knee joint
* Inflammatory and Infectious knee conditions (RA, gout, psoriatic arthritis)
* Balance problem
* Any recent surgical intervention of knee joint or those who had undergone arthroplasty
* Surgeries in hip or knee
* Tumors/malignancy of bone

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Western Ontario & Mc-master Osteoarthritis Index | 12 weeks
  The WOMAC takes approximately 12 minutes to complete, and can be taken on paper, over the telephone or computer. Both the computerized and the mobile versions of the test have been found to be comparable to the paper form, with no significant difference.
  The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
Time Up & Go Test | 12 weeks
  An older adult who takes ≥12 seconds to complete the TUG is at risk for falling.
  Cut of scores indicating risk of falls by Population (in seconds) Community dwelling adults - 13.5 Older stroke patients - 14 Frail elderly - 32.6 LE amputees - 19 PD - 11.5 Hip OA - 10 - Vestibular disorders - 11.1 Cut-off times to classify subjects as high risk for falling vary based on the study and participants.
Numeric Pain Rating Scale | 12 weeks
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults,including those with chronic pain due to rheumatic diseases.
  0 means no pain and 10 means the worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hashim, PPDPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goh SL, Persson MSM, Stocks J, Hou Y, Welton NJ, Lin J, Hall MC, Doherty M, Zhang W. Relative Efficacy of Different Exercises for Pain, Function, Performance and Quality of Life in Knee and Hip Osteoarthritis: Systematic Review and Network Meta-Analysis. Sports Med. 2019 May;49(5):743-761. doi: 10.1007/s40279-019-01082-0. PMID 30830561
- [Background] Gondhalekar GA, Deo MV. Retrowalking as an adjunct to conventional treatment versus conventional treatment alone on pain and disability in patients with acute exacerbation of chronic knee osteoarthritis: a randomized clinical trial. N Am J Med Sci. 2013 Feb;5(2):108-12. doi: 10.4103/1947-2714.107527. PMID 23641371
- [Background] Jeong HS, Lee SC, Jee H, Song JB, Chang HS, Lee SY. Proprioceptive Training and Outcomes of Patients With Knee Osteoarthritis: A Meta-Analysis of Randomized Controlled Trials. J Athl Train. 2019 Apr;54(4):418-428. doi: 10.4085/1062-6050-329-17. Epub 2019 Apr 17. PMID 30995119
- [Background] Black DW. Treatment of knee arthrofibrosis and quadriceps insufficiency after patellar tendon repair: a case report including use of the graston technique. Int J Ther Massage Bodywork. 2010 Jun 23;3(2):14-21. PMID 21589706
- [Background] Chen ZH, Ye XL, Chen WJ, Chen GQ, Wu JT, Wu H, Xu XM. Effectiveness of backward walking for people affected by stroke: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2020 Jul 2;99(27):e20731. doi: 10.1097/MD.0000000000020731. PMID 32629648